CLINICAL TRIAL: NCT02194218
Title: An Open-label, Randomised, Single Dose, Parallel-group Phase I Study to Investigate the Pharmacokinetic Properties of 200 mg Nevirapine Extended Release Tablets When Administered Orally as 2x100 mg Tablets or as 4x50 mg Tablets in Healthy Male Volunteers
Brief Title: Pharmacokinetic Properties of Nevirapine Extended Release Tablets When Administered Orally in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1100.1531
Record Dates: First submitted 2014-07-17; First posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Nevirapine

ARMS (2):
- Nevirapine XR 4 doses (Experimental)
  Interventions: Drug: Nevirapine, low dose
- Nevirapine XR 2 doses (Active Comparator)
  Interventions: Drug: Nevirapine, high dose

INTERVENTIONS:
Drug: Nevirapine, low dose — 50 mg
  Arms: Nevirapine XR 4 doses
Drug: Nevirapine, high dose — 100 mg
  Arms: Nevirapine XR 2 doses

SUMMARY:
Study to determine the pharmacokinetic properties of 200 mg nevirapine (NVP) administered as 4 x 50 mg extended release (XR) tablets in a single dose and to establish the bioequivalence of this formulation compared to 200 mg NVP administered as 2 x 100 mg XR tablets in a single dose

ELIGIBILITY:
Inclusion Criteria:

* Healthy male according to the following criteria based upon a complete medical history, including the physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead electrocardiogram (ECG), clinical laboratory; values within normal ranges or deviating from normal without clinical relevance as considered by the investigator
* Age ≥21 and Age ≤50 years
* Body Mass Index (BMI) ≥18.5 and BMI ≤29.9 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with Good clinical practice (GCP) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders of clinical relevance
* Surgery of the gastrointestinal tract (except appendectomy and herniotomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Previous intake of Nevirapine
* Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 30 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 144 hours post-dose
Maximum measured concentration of the analyte in plasma (Cmax) | up to 144 hours post-dose

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point (AUC0-tz) | up to 144 hours post-dose
Time from dosing to the maximum concentration of the analyte in plasma (tmax) | up to 144 hours post-dose
Terminal rate constant in plasma (λz) | up to 144 hours post-dose
Terminal half-life of the analyte in plasma (t1/2) | up to 144 hours post-dose
Mean residence time of the analyte in the body after po administration (MRTpo) | up to 144 hours post-dose
Apparent clearance of the analyte in the plasma after extravascular administration (CL/F) | up to 144 hours post-dose
Apparent volume of distribution during the terminal phase λz following an extravascular dose (Vz/F) | up to 144 hours post-dose
Absorption rate constant (ka) | up to 144 hours post-dose
Number of patients with adverse events | up to 35 days
Assessment of tolerability by investigator on a 4-point scale | within 8 days after last trial procedure